CLINICAL TRIAL: NCT06250153
Title: In-Person Versus Text/Telephone Screening, Brief Intervention and Referral to Treatment in Primary Care
Brief Title: TAU vs m-SBIRT in Primary Care
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: funding
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Pro00133783
Record Dates: First submitted 2024-01-27; First posted 2024-02-08 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Substance Use Disorders
Keywords: Substance Use Disorders; Social Determinants of Health; Screening, Brief Intervention, Referral to Treatment (SBIRT); Telehealth; Mobile SBIRT (m-SBIRT); Primary Care
MeSH Terms: conditions — Substance-Related Disorders | interventions — Crisis Intervention

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (No Intervention): This group will receive routine substance use screening questions during their in-person primary care visit as part of standard of care.
- m-SBIRT (mobile-Screening, Brief Intervention, and Referral to Treatment) (Experimental): This group will receive a mobile phone text message based substance use screening (questions used in standard of care) with immediate automated feedback, paired with remote care coordination and, if appropriate, referral to substance use disorder (SUD) treatment.
  Interventions: Behavioral: m-SBIRT (mobile-Screening, Brief Intervention, and Referral to Treatment)

INTERVENTIONS:
Behavioral: m-SBIRT (mobile-Screening, Brief Intervention, and Referral to Treatment) — M-SBIRT is a mobile phone-based program designed to enhance delivery of Screening, Brief Intervention, and Referral to Treatment (SBIRT), an evidence-based approach for mental health and substance use screening and treatment. The program utilizes mobile phone text message-based screenings with immediate automated feedback, paired with remote care coordination and, if appropriate, referral to substance use disorder treatment services.
  Arms: m-SBIRT (mobile-Screening, Brief Intervention, and Referral to Treatment)

SUMMARY:
The goal of this research is to leverage technology in primary care clinics to improve screening, brief intervention and referral to Substance Use Disorder (SUD) treatment, and treatment attendance by comparing

1. a text message-based screening, phone-based brief intervention, and referral to treatment by a remote care coordinator (m-SBIRT; intervention arm), versus
2. evidence-based, in-person Screening, Brief Intervention, and Referral to Treatment (SBIRT; Treatment As Usual (TAU); control arm).

Primary Aim is to compare the efficacy of m-SBIRT to TAU in positive screens for substance use. Secondary Aim is to compare m-SBIRT to TAU on Substance Use Treatment Attendance.

DETAILED DESCRIPTION:
This research study is looking at the use of technology in primary care clinics and seeing if it improves screening, brief intervention and referral to Substance Use Disorder (SUD) treatment, and attendance to treatment. To do so the study, Investigators will be comparing a text message based substance use screening and treatment program, called Mobile Screening, Brief intervention, and Referral to Treatment (m-SBIRT) to standard of care Screening, Brief Intervention and Referral Treatment which traditionally takes place in-person. Patients at the MUSC Bee Street Primary Care Clinic between the ages of 18-75 may be eligible.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* Attended a primary care visit at the MUSC Family Medicine clinic on Bee St
* English fluency
* Owner of a cell phone with SMS text-message based capability
* Access to WIFI
* A device to allow audio and video teleconferencing if completing informed consent remotely
* Able to provide informed consent.

Exclusion Criteria:

- None

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Positive screens for substance use | Immediately following screening.
  A positive screen is defined as positive endorsement of substance use (alcohol, drugs, tobacco, etc) within the questionnaire. We will compare rates of positive screens for substance use in individuals assigned to m-SBIRT compared to TAU.
Change in treatment attendance | Within one month of referral to treatment.
  Treatment attendance is defined as attending one or more visits to address substance use concerns within one month of referral. We will compare rates of treatment attendance of individuals assigned to m-SBIRT compared to TAU.

CONTACTS AND LOCATIONS:
Overall Officials: Constance Guille, MD, Principal Investigator — Professor-Faculty